CLINICAL TRIAL: NCT07153523
Title: Effect of High Intensity Interval Training Versus Conservative Treatment on Strength, Endurance and Flexibility of Undergraduate Physical Therapy Students
Brief Title: Effect of High Intensity Interval Training on Strength, Endurance and Flexibility
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Health Sciences Lahore (Other)
Responsible Party: Principal Investigator, Wajeeha Mahmood, Dr Wajeeha Mahmood(PT), University of Health Sciences Lahore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UHS/DPS-25/1205
Record Dates: First submitted 2025-08-25; First posted 2025-09-04 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: High Intensity Interval Training
Keywords: high intensity interval training
MeSH Terms: interventions — High-Intensity Interval Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental arm (Experimental): High intensity interval training
  Interventions: Other: High intensity interval training
- Control arm (Active Comparator): routine physical therapy
  Interventions: Other: Routine physical therapy

INTERVENTIONS:
Other: High intensity interval training — High intensity interval training provides time efficient benefits for strength and endurance training. It comprises of high burst training with rest periods. For experimental group HIIT training will be applied comprising of burpees, squats, arm walking and lunges. The exercise will be given 3 times/ week for 4 weeks. For standardization experimental group will receive 10 minutes of warm up and cool down period comprising of stretching exercises
  Arms: Experimental arm
Other: Routine physical therapy — For control group routine physical therapy will be applied for strength training using weights and running drills for endurance training. The exercise will be given 3 times/ week for 4 weeks. For standardization control group will receive 10 minutes of warm up and cool down period comprising of stretching exercises
  Arms: Control arm

SUMMARY:
Strength and endurance are essential components for physical fitness of any individual. High intensity interval training provides time efficient benefits for strength and endurance training. Physical Therapy professionals and students need physical fitness for effective clinical performance of patients. There is limited research regarding physical performance of physical therapists itself

DETAILED DESCRIPTION:
Physical fitness is defined as capacity of doing physical activity using muscular efforts, resulting in energy expenditure. It is dependent upon body composition, muscle strength, endurance and flexibility of person. Pre assessment of strength, endurance and flexibility among physical therapy students will measure their physical fitness and findings from High intensity interval training (HIIT) will help further clinicians for designing fitness program to enhance physical abilities of future physical therapists. This study will address the gap by finding effects of HIIT that would help to improve fitness level of physical therapy students and influence exercise prescription.

Objective: To determine effects of high intensity interval training versus conservative treatment for strength, endurance and flexibility of undergraduate physical therapy students

ELIGIBILITY:
Inclusion Criteria:

* Undergraduate physical therapy students aged 18-24 years.
* Both genders male and female
* DPT students from 1st to final year

Exclusion Criteria:

* Students with musculoskeletal pain and injuries.
* Any neurological and cardiovascular restrictions.
* Any trauma like fracture.
* Surgical limitation of range of motion.
* Any systemic disease.
* Malignant or benign Tumor.
* Students who are athletes or doing regular exercise

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Estimated)
Dates: Start 2025-08-21 (Actual); Primary Completion 2025-11-15 (Estimated); Study Completion 2025-11-20 (Estimated)

PRIMARY OUTCOMES:
Strength | From enrollment to the end of treatment at 4 weeks
  The grip strength will be measured using Hand Held Dynamometer (model). Lower limb strength will be measured through vertical jump test
Muscle endurance | From enrollment to the end of treatment at 4 weeks
  The sit-up test will be used to assess muscular endurance
Flexibility | From enrollment to the end of treatment at 4 weeks
  The flexibility will be assessed using sit and reach test

CONTACTS AND LOCATIONS:
Locations (1):
- Dr Wajeeha Mahmood (PT), Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No